CLINICAL TRIAL: NCT01043484
Title: Phase II Randomized Study to Compare Capecitabine + Bevacizumab Concomitantly With Radiotherapy Versus Capecitabine Concomitantly With Radiotherapy, as Neoadjuvant Treatment for Patients With Localized and Resectable Rectal Cancer
Brief Title: Safety and Efficacy Study to Compare Capecitabine + Bevacizumab Versus Capecitabine, Concomitantly With Radiotherapy as Neoadjuvant Treatment for Patients With Localized and Resectable Rectal Cancer
Acronym: AVAXEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-08-05; EudraCT: 2009-010192-24
Record Dates: First submitted 2009-12-30; First posted 2010-01-06 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Rectal Cancer
Keywords: Resectable rectal cancer; Radiotherapy; Bevacizumab; Capecitabine
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Bevacizumab + Capecitabine + Radiotherapy
  Interventions: Drug: Bevacizumab + Capecitabine + Radiotherapy
- B (Active Comparator): Capecitabine + Radiotherapy
  Interventions: Drug: Capecitabine + Radiotherapy

INTERVENTIONS:
Drug: Bevacizumab + Capecitabine + Radiotherapy — Bevacizumab (5 mg/kg; days 1, 15 and 29) Capecitabine (825 mg/m2/12h, 5 days/w) Radiotherapy (45 Gy in sessions of 1.8 Gy 5 times/w for 5 weeks)
  Arms: A
Drug: Capecitabine + Radiotherapy — Capecitabine (825 mg/m2/12h, 5 days/w) and Radiotherapy (45 Gy in sessions of 1.8 Gy 5 times/w for 5 weeks)
  Arms: B

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the combination of capecitabine + bevacizumab concomitantly with radiotherapy versus capecitabine concomitantly with radiotherapy, as neoadjuvant treatment for patients with localized and resectable rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* ECOG ≤ 1
* Histologically confirmed carcinoma of the rectum
* Localized and resectable rectal cancer
* No metastatic disease
* Measurable disease
* Life expectancy more than 4 months
* Non prior treatment for rectal cancer
* Adequate haematological function: leu ≥ 4x 109 /l, Hb ≥10 gr/dl, neutropils≥ 1,5 x 109 /l and platelets ≥100 x 109 /l
* Adequate renal function: creatinine ≤ 106 umol/l or calculated creatinine clearance > 50 mL/min
* Adequate liver function: AST, ALT and alkaline phosphatase ≤2.5 x UL, bilirubin ≤1.5 x UL
* Adequate nutritional weight loss <10% of regular weight and albumin ≥ 35 g/l

Exclusion Criteria:

* Unresectable rectal cancer
* Past or current history (within the last 5 years prior to treatment start) of other malignancies.
* Patients of childbearing potential not willing to use effective means of contraception.
* Clinically significant cardiovascular disease
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome or inability to take oral medication.
* Patients subjected to organ allografts who require immunosuppressive treatment.
* Severe, non-cicatrized osseous fractures, wounds or ulcers.
* Indications of hemorrhagic diathesis or coagulopathy.
* Severe, uncontrolled intercurrent infections or other severe, uncontrolled concomitant diseases.
* History of unexpected severe reactions to treatment with fluoropyrimidines or known deficiency dihydropyrimidine dehydrogenase deficiency (DPD).
* Patients subjected to a major surgical procedure, open biopsy or who have had significant traumatic lesions within the 28 days prior to beginning the treatment of the study or in whom it is foreseen that a major surgical procedure will be necessary during the course of the study; fine-needle aspiration within the 7 days prior to beginning the treatment of the study.
* Current or recent use (within the 10 days prior to beginning the treatment of the study) of oral or parenteral anticoagulants at complete doses or thrombolytic agents. The use of low doses of warfarin is allowed, with an International Normalized Ratio [INR] of < 1.5.
* Daily chronic treatment with high doses of aspirin (> 325 mg/day) or non-steroid anti-inflammatory medications (which inhibit the platelet function at doses used for treating chronic inflammatory diseases).
* Patients who have received any drug or agent/procedure under research, i.e., who have participated in another clinical trial during the 4 weeks prior to beginning the treatment with the medications of the study
* Any psychological, familiar conditions suggesting that the patient will not be able to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Rate complete pathologic responses | 17 months

SECONDARY OUTCOMES:
Disease free survival at 3 and 5 years | 78 months
Rate of local and distant recurrence at 3 and 5 years | 78 months
Overall survival at 3 and 5 years | 78 months
R0 resection rate. | 17 months
Adverse events | 17 months
Rate of surgery complications | 17 months
Molecular predictive markers: changes in angiogenic parameters, vascular endothelial growth factor (VEGF), vascular endothelial growth factor receptors, microvessel quantification and angiopoietin-2 (Ang-2) | 17 months
Rate of sphincter preservation | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Salazar, Study Chair — Institut Català d´Oncologia (ICO) L'Hospitalet. Barcelona. Spain; Cristina Grávalos, Study Chair — Hospital 12 Octubre. Madrid. Spain; Sebastiano Biondo, Study Chair — Hospital Universitario de Bellvitge.Barcelona. Spain; Amalia Palacios, Study Chair — Hospital Universitario Reina Sofía. Córdoba. Spain
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Salazar R, Capdevila J, Manzano JL, Pericay C, Martinez-Villacampa M, Lopez C, Losa F, Safont MJ, Gomez-Espana A, Alonso-Orduna V, Escudero P, Gallego J, Garcia-Paredes B, Palacios A, Biondo S, Gravalos C, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD). Phase II randomized trial of capecitabine with bevacizumab and external beam radiation therapy as preoperative treatment for patients with resectable locally advanced rectal adenocarcinoma: long term results. BMC Cancer. 2020 Nov 27;20(1):1164. doi: 10.1186/s12885-020-07661-z. PMID 33246428
- [Derived] Salazar R, Capdevila J, Laquente B, Manzano JL, Pericay C, Villacampa MM, Lopez C, Losa F, Safont MJ, Gomez A, Alonso V, Escudero P, Gallego J, Sastre J, Gravalos C, Biondo S, Palacios A, Aranda E. A randomized phase II study of capecitabine-based chemoradiation with or without bevacizumab in resectable locally advanced rectal cancer: clinical and biological features. BMC Cancer. 2015 Feb 26;15:60. doi: 10.1186/s12885-015-1053-z. PMID 25886378
- See also: Related Info — http://www.ttdgroup.org